CLINICAL TRIAL: NCT04780542
Title: Computerized Detection and Internet-based Treatment of Common Mental Disorders Among College Students in Two Latin American LMICs
Brief Title: Internet-delivered Cognitive Behavioral Treatment of Depression and Anxiety in Latin American College Students
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Psiquiatría Dr. Ramón de la Fuente (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Corina Benjet, Principal Investigator, Instituto Nacional de Psiquiatría Dr. Ramón de la Fuente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EP20142; R01MH120648-01A1 (NIH)
Record Dates: First submitted 2021-02-28; First posted 2021-03-03 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Major Depressive Disorder; Generalized Anxiety Disorder
Keywords: iCBT; Latin America; College Students; Depression; Anxiety
MeSH Terms: conditions — Depressive Disorder, Major; Generalized Anxiety Disorder; Depression; Anxiety Disorders

STUDY DESIGN:
Masking Description: Participant recruiters will be blinded to the participant's intended treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinician-Guided iCBT (Experimental): Both help-seeking students recruited from university clinics and non-help-seeking students recruited from needs assessment survey and outreach will receive internet delivered cognitive behavioral therapy guided by clinicians
  Interventions: Behavioral: Yo Puedo Sentirme Bien- Clinician-Guided version
- Self-guided iCBT (Active Comparator): Help-seeking students recruited from university clinics will receive self-guided internet delivered cognitive behavioral therapy while on waitlist. Non-help seeking students recruited from needs assessment survey and outreach will receive the self-guided version of internet delivered cognitive behavioral therapy.
  Interventions: Behavioral: Yo Puedo Sentirme Bien- Self-Guided version

INTERVENTIONS:
Behavioral: Yo Puedo Sentirme Bien- Clinician-Guided version — Internet delivered Cognitive Behavioral Therapy- Guided version
  Arms: Clinician-Guided iCBT
Behavioral: Yo Puedo Sentirme Bien- Self-Guided version — Internet delivered Cognitive Behavioral Therapy- Self-Guided version
  Arms: Self-guided iCBT

SUMMARY:
The aim is to evaluate short term and longer term treatment effects of internet-delivered cognitive behavioral therapy compared to treatment as usual for college students with anxiety and/or depression in low-middle income countries of Latin America.

DETAILED DESCRIPTION:
This study is designed to detect, engage, and experimentally evaluate the effects of internet-based cognitive behavior therapy (e-CBT) to treat college students in two Latin American low-middle income countries (LMICs; Colombia and Mexico) with major depressive disorder and/or generalized anxiety disorder, with or without other comorbid common mental disorders (CMDs). Detection and engagement will be based on inexpensive internet-based recruitment and administration of self-report surveys. The intervention will be based on inexpensive e-CBT to address the low resources in LMICs. The study builds on prior research by collaborators in the WHO World Mental Health (WMH) survey consortium and WMH International College Study (WMH-ICS) initiative documenting high prevalence, impairment, and unmet need for treatment of CMDs among college students around the world and significant effects of e-CBT in treating these disorders in high income countries.

First, the investigators will carry out a pragmatic clinical trial with students seeking treatment for CMDs at student clinics in universities in Colombia and Mexico. Students on waitlists for student clinic services will be offered a possibility of receiving guided or self-guided e-CBT immediately while staying on the list. 33% of the students with CMD who express interest will be randomized to guided e-CBT, another 33% to self-guided e-CBT, and the remaining 33% to treatment as usual (TAU), where the latter is defined as remaining on the waiting list. Short-term aggregate intervention effects will be assessed 90 days after randomization and longer-term effects 12 months after randomization. The investigators will then use ensemble machine learning methods to predict heterogeneity of treatment effects of e-CBT versus TAU and develop a precision treatment rule (PTR) to predict which students will respond best to which intervention. A SMART design will then be implemented in which 50% of a second cohort of students from the same sample frame (i.e., students seeking treatment for CMDs at student clinics in the participating universities) will be randomized to the treatment arm predicted to be optimal by the PTR and the other 50% to randomization across arms. Based on the findings from the first pragmatic trial, none of the students were optimized by TAU. Therefore for the next cohort of students they will be randomized only to two arms, guided and unguided. Additionally, the investigators will use outreach to recruit students into the trial who might not otherwise seek treatment from student clinics. Two procedures will be used here. In the first, students will be recruited from annual WMH-ICS internet-based mental health needs assessment surveys that will be carried out with a probability sample of students to estimate unmet need for treatment and barriers to treatment. Students who respond to these surveys and meet inclusion criteria and are not in treatment will be randomized to guided e-CBT, self-guided e-CBT, and treatment as usual (only in first pragmatic trial) in student clinics to determine if access to guided and self-guided e-CBT reduces the unmet need for treatment among students with CMDs who fail to seek treatment at student health clinics. The second will expand recruitment by sending emails to random subsamples of students notifying them of the availability of the internet-based interventions and inviting them to participate in a trial. Students that respond to this announcement will then be recruited and randomized into the same three arms as among students that participated in the annual WMH-ICS survey.

ELIGIBILITY:
Inclusion Criteria:

At least 18 years of age, screens positive for major depressive disorder and/or generalized anxiety disorder, student enrolled in one of the participating universities

Exclusion Criteria:

Screens positive for bipolar disorder, screens positive for psychosis, active suicidality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | 90 days
  Self-report measure of depressive symptoms in the prior 2 weeks. Scores range from 0 to 27 with higher scores representing greater depressive symptomatology.
Generalized Anxiety Disorder-7 (GAD-7) | 90 days
  Self-report measure of anxiety symptoms in the prior 2 weeks. Scores range from 0 to 21 with higher scores representing greater anxiety.
Patient Health Questionnaire-9 (PHQ-9) | 12 months
  Self-report measure of depressive symptoms in the prior 2 weeks. Scores range from 0 to 27 with higher scores representing greater depressive symptomatology.
Generalized Anxiety Disorder-7 (GAD-7) | 12 months
  Self-report measure of anxiety symptoms in the prior 2 weeks. Scores range from 0 to 21 with higher scores representing greater anxiety.

SECONDARY OUTCOMES:
(Army STARRS) Role impairment | 90 days
  Self-report measure of impairment due to mental health in four life areas in the prior 2 weeks. Scores in each area range from 0 to 10 with higher scores reflecting greater impairment.
(Army STARRS) Role impairment | 12 months
  Self-report measure of impairment due to mental health in four life areas in the prior 2 weeks. Scores in each area range from 0 to 10 with higher scores reflecting greater impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Corina Benjet, PhD, Principal Investigator — Instituto Nacional de Psiquiatría
Locations (8):
- Colombia (4):
  - Universidad Nacional de Colombia, Bogotá
  - Universidad Cooperativa de Colombia, Medellín
  - Fundación Universitaria del Area Andina, Valledupar
  - Universidad Popular de Cesar, Valledupar
- Mexico (4):
  - Universidad Autonoma de Baja California, Ensenada
  - Universidad la Salle, León
  - Universidad Autonoma Metropolitana, Mexico City
  - Universidad Nacional Autonoma de México, Mexico City

IPD SHARING:
Plan to Share IPD: Yes
First, we will document and make available all imputations, weights, and constructed variables used in our analyses. Second, we will host a project webinars to present an overview of the data and answer questions. The webinars will be widely advertised in list serves, including any such sites recommended by NIMH, as well as to NIH training programs. An English version of the webinars will be hosted by the US collaborators. A Spanish version will be hosted by the Mexican collaborators. Third, we will set up and man a project Q&A web site in which public users can ask questions and get answers about issues involved in working with the data. Again, the site will be both in English and Spanish. Fourth, we will gather up written versions of all questions asked by public users along with our written response (including any documentation or computer files sent along with these answers) and post these on the website in both English and Spanish as reference documents for future public users.
Supporting Information: Study Protocol, CSR
Time Frame: Data will become available in Year 5, once trials are concluded
Access Criteria: By written request

REFERENCES:
- [Derived] Benjet C, Zainal NH, Albor Y, Alvis-Barranco L, Carrasco Tapia N, Contreras-Ibanez CC, Cortes-Morelos J, Cudris-Torres L, de la Pena FR, Gonzalez N, Gutierrez-Garcia RA, Vargas-Contreras E, Medina-Mora ME, Patino P, Gildea SM, Kennedy CJ, Luedtke A, Sampson NA, Petukhova MV, Zubizarreta JR, Cuijpers P, Kazdin AE, Kessler RC. The Effect of Predicted Compliance With a Web-Based Intervention for Anxiety and Depression Among Latin American University Students: Randomized Controlled Trial. JMIR Ment Health. 2025 Feb 28;12:e64251. doi: 10.2196/64251. PMID 40053727
- [Derived] Benjet C, Albor Y, Alvis-Barranco L, Contreras-Ibanez CC, Cuartas G, Cudris-Torres L, Gonzalez N, Cortes-Morelos J, Gutierrez-Garcia RA, Medina-Mora ME, Patino P, Vargas-Contreras E, Cuijpers P, Gildea SM, Kazdin AE, Kennedy CJ, Luedtke A, Sampson NA, Petukhova MV, Zainal NH, Kessler RC. Internet-delivered cognitive behavior therapy versus treatment as usual for anxiety and depression among Latin American university students: A randomized clinical trial. J Consult Clin Psychol. 2023 Dec;91(12):694-707. doi: 10.1037/ccp0000846. PMID 38032621
- [Derived] Benjet C, Zainal NH, Albor Y, Alvis-Barranco L, Carrasco-Tapias N, Contreras-Ibanez CC, Cudris-Torres L, de la Pena FR, Gonzalez N, Guerrero-Lopez JB, Gutierrez-Garcia RA, Jimenez-Perez AL, Medina-Mora ME, Patino P, Cuijpers P, Gildea SM, Kazdin AE, Kennedy CJ, Luedtke A, Sampson NA, Petukhova MV, Kessler RC. A Precision Treatment Model for Internet-Delivered Cognitive Behavioral Therapy for Anxiety and Depression Among University Students: A Secondary Analysis of a Randomized Clinical Trial. JAMA Psychiatry. 2023 Aug 1;80(8):768-777. doi: 10.1001/jamapsychiatry.2023.1675. PMID 37285133
- [Derived] Benjet C, Kessler RC, Kazdin AE, Cuijpers P, Albor Y, Carrasco Tapias N, Contreras-Ibanez CC, Duran Gonzalez MS, Gildea SM, Gonzalez N, Guerrero Lopez JB, Luedtke A, Medina-Mora ME, Palacios J, Richards D, Salamanca-Sanabria A, Sampson NA. Study protocol for pragmatic trials of Internet-delivered guided and unguided cognitive behavior therapy for treating depression and anxiety in university students of two Latin American countries: the Yo Puedo Sentirme Bien study. Trials. 2022 Jun 2;23(1):450. doi: 10.1186/s13063-022-06255-3. PMID 35658942